CLINICAL TRIAL: NCT02225327
Title: Immunogenicity and Safety of MF59-adjuvanted Trivalent Influenza Vaccine (Fluad) and 23-valent Pneumococcal Polysaccharide Vaccine (PPV23) in the Elderly: Single Versus Concomitant Vaccination
Brief Title: MF59-adjuvanted Influenza Vaccine and 23-valent Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Hee Jin Cheong, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLUADPPV23
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Influenza, Human; Pneumococcal Infections
MeSH Terms: conditions — Influenza, Human; Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fluad alone (Active Comparator): 56 Fluad recipients: one vaccine injection administered on Day 0
  Interventions: Biological: Fluad alone
- Fluad and PPV23 on the different arms (Active Comparator): 56 concomitant Fluad-PPV23 recipients on the different arms: one dose of each vaccine administered on Day 0
  Interventions: Biological: Fluad and PPV23 on the different arms
- Fluad and PPV23 on the same arm (Active Comparator): 56 concomitant Fluad-PPV23 recipients on the same arm with 1 inch distance: one dose of each vaccine administered on Day 0
  Interventions: Biological: Fluad and PPV23 on the same arm
- PPV23 alone (Active Comparator): 56 PPV23 recipients: one vaccine injection administered on Day 0
  Interventions: Biological: PPV23 alone

INTERVENTIONS:
Biological: Fluad alone — Fluad
  Arms: Fluad alone
Biological: Fluad and PPV23 on the different arms — Fluad and Prodiax
  Arms: Fluad and PPV23 on the different arms
Biological: Fluad and PPV23 on the same arm — Fluad and Prodiax
  Arms: Fluad and PPV23 on the same arm
Biological: PPV23 alone — Prodiax
  Arms: PPV23 alone

SUMMARY:
Similar to children, adults frequently visit outpatient clinics to get two or more kinds of vaccines at the same time: pneumococcal vaccine, influenza vaccine, Td (diphtheria and tetanus) vaccine, HPV (human papilloma virus) vaccine, meningococcal vaccine, zoster vaccine, etc. This study is intended to evaluate the immunogenicity and safety of concomitant administration of 23-valent pneumococcal polysaccharide vaccine (PPV23, Prodiax) and MF59 adjuvanted trivalent influenza vaccine in the elderly subjects aged ≥65 years.

DETAILED DESCRIPTION:
During influenza season, concomitant influenza and pneumococcal vaccination would be an effective strategy to enhance pneumococcal vaccine coverage rate in high-risk adults. However, the immunogenicity and safety of concomitant vaccination need to be further investigated. There is data on immunogenicity and safety after concomitant administration of pneumococcal polysaccharide vaccine (PPV) and unadjuvanted influenza vaccine; no interference was noted between two vaccines. However, there are no data for MF59 adjuvanted influenza vaccine with pneumococcal vaccine. MF59 only locally reacts for immune response, so immunogenicity should be assessed for both vaccines injected in same arm versus different arms.

This study is intended to evaluate the immunogenicity and safety of concomitant MF59-adjuvanted trivalent influenza vaccine (MF59-aTIV, Fluad) and 23-valent pneumococcal polysaccharide vaccine (PPV23, Prodiax) vaccination in the elderly subjects aged ≥65 years. Healthy elderly subjects (N = 424) are randomized in a 1:1:1:1 ratio to receive MF59-aTIV alone (group 1), MF59-aTIV +PPV23 at different arm (group 2), MF59-aTIV +PPV23 at same arm (group 3) or PPV23 alone (group 4).

Hemagglutination inhibition (HI) assay and multiplex opsono-phagocytic killing assay (MOPA) will be used to compare the immunogenicity of each vaccine after single or concomitant vaccination at pre-vaccination and 1 month post-vaccination. MOPA will be taken for four serotypes (5, 6B, 18C and 19A).

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years of age who are eligible for the study vaccines;
* Who have given written informed consent at the time of enrollment);
* Those who are available for all the visits scheduled in the study;
* Subjects In good health as determined by medical history, physical examination and clinical judgment of the investigator

Exclusion Criteria:

* History of egg allergy
* History of influenza vaccination in previous 6 months
* History of any pneumococcal vaccination
* Documented S. pneumonia infection in the previous 5 years
* Chemotherapy for malignancy within the past 30 days
* High-dose systemic steroid (prednisone ≥0.5 mg/kg/day) in the past 30 days
* Receipt of blood product within 6 months before enrollment
* Significant acute or chronic infection within the previous 7 days or fever within the previous day
* Any serious chronic or progressive disease
* Any condition that might interfere with the study results.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates (A/H1N1, A/H3N2, and B) | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination)
  a post-vaccination titer ≥1:40 in subjects with a pre-vaccination titer of <1:10 or a ≥4-fold titer increase in subjects with a pre-vaccination titer of ≥1:10

SECONDARY OUTCOMES:
Seroprotection rates (A/H1N1, A/H3N2, and B) | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination).
  Percentage of subjects with a post-vaccination titer ≥1:40
GMT folds (A/H1N1, A/H3N2, and B) | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination.
  GMT-fold change: GMT ratio of the post-vaccination titer to pre-vaccination titer
Opsonophagocytic assay (OPA) titers for four serotypes of PPV23 (serotypes 5, 6B, 18C and 19A) | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination).
  OPA geometric mean titers for four PPV23 serotypes with corresponding 2-sided 95% confidence intervals will be compared between groups receiving PPV23: MF59-adjuvanted TIV + PPV23 at different arm, MF59-adjuvanted TIV + PPV23 at same arm and PPV23 alone.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, MD, PhD, Principal Investigator — Korea University Guro Hospital; Joon Young Song, MD, PhD, Study Director — Korea University Guro Hospital

REFERENCES:
- [Derived] Song JY, Cheong HJ, Tsai TF, Chang HA, Choi MJ, Jeon JH, Kang SH, Jeong EJ, Noh JY, Kim WJ. Immunogenicity and safety of concomitant MF59-adjuvanted influenza vaccine and 23-valent pneumococcal polysaccharide vaccine administration in older adults. Vaccine. 2015 Aug 26;33(36):4647-52. doi: 10.1016/j.vaccine.2015.05.003. Epub 2015 May 14. PMID 25980426